CLINICAL TRIAL: NCT00403949
Title: A 6-week, Vehicle-controlled, Randomized, Double-blind, Parallel-group Multicenter Pilot Study of the Efficacy and Safety of Azelaic Acid (AzA) 15% Gel in the Topical Treatment of Mild to Moderate Perioral Dermatitis
Brief Title: A Study of Azelaic Acid (AzA) 15% in Topical Treatment of Mild to Moderate Perioral Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1400418; 2006-002471-40 (EudraCT Number)
Record Dates: First submitted 2006-11-23; First posted 2006-11-27 (Estimated); Last update posted 2023-06-09 (Actual); Status verified 2015-02

CONDITIONS: Perioral Dermatitis
MeSH Terms: conditions — Dermatitis, Perioral | interventions — azelaic acid; Gels

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Azelaic acid 15% Gel (Active Comparator): Azelaic acid 15%
  Interventions: Drug: Azelaic acid 15% gel
- Placebo (Placebo Comparator): Non-active base from Azelaic acid 15% gel
  Interventions: Drug: Non-active base from azelaic acid 15% gel

INTERVENTIONS:
Drug: Azelaic acid 15% gel — gel, applied once daily, for 6 weeks
  Arms: Azelaic acid 15% Gel
Drug: Non-active base from azelaic acid 15% gel — gel, apply once daily for six weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the efficacy and safety of AzA 15% Gel in the treatment of mild to moderate perioral dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of mild to moderate perioral dermatitis as diagnosed by the physician
* Investigator's Global Assessment (IGA) score at baseline of 2 or 3 (on scale from 0 to 4)
* 8 to 50 facial inflammatory lesions (papules, papulopustules, papulovesicles)

Exclusion Criteria:

* History of atopic dermatitis of the face
* Granulomatous perioral dermatitis
* Facial acne, rosacea, facial demodicosis
* Seborrheic dermatitis of the nasolabial fold, Lupus erythematosus
* The use of topical or systemic medications that could affect the course of treatment and/or evaluation
* Severe diseases likely to interfere with the conduct / planned termination of the study (e.g. cancer, cardiac infarct, unstable angina pectoris, uncontrolled diabetes)
* Use of fluorinated toothpaste
* Planned exposure to artificial or intensive natural UV light of the test area throughout the course of the study
* Use / planned use of cosmetic products (e.g. creams, moisturizers, make-up, fatty lipstick) in the test area during the course of the study
* History of or suspected hypersensitivity to any ingredient of the study drugs
* Participation in another clinical study 4 weeks prior to and/or during the conduct of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2006-11; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
The sum score derived from the most important signs and symptoms of perioral dermatitis | Measurements and observations during the course of the study

SECONDARY OUTCOMES:
Intensity of single signs and symptoms | Measured at scheduled visits during the course of the study
Safety outcomes measures will be all adverse events reported by the patients or observed by the investigator | Safety parameters recorded at scheduled visits during the course of the study

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (4):
- Germany (4):
  - Berlin
  - Dülmen
  - Essen
  - Recklinghausen